CLINICAL TRIAL: NCT02505139
Title: Using Circulating Tumor Cells to Diagnose and Predict Prognosis in Metastatic Nasopharyngeal Carcinoma Patients
Brief Title: The Value of Diagnosis and Outcome Prediction in CTC for Metastatic NPC Patients
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Prof., Sun Yat-sen University
Other Study IDs: SYSUCCCTC
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: nasopharyngeal carcinoma; distant metastasis; circulating tumor cells; outcome prediction
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The blood after separation and purification along with or without CTC.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study Group
  Interventions: Other: the number of circulating tumor cells

INTERVENTIONS:
Other: the number of circulating tumor cells

SUMMARY:
A circulating tumor cell (CTC) count is an established prognostic factor in some malignancies such as metastatic breast cancer. However, the value of CTC in diagnosis and outcome prediction of metastatic nasopharyngeal carcinoma (mNPC) patients is not unknown. Through the observational prospective clinical trial, sensitivity, specificity, positive and negative predictive values of CTC in diagnosis of mNPC patients will be gained. Further, the value of CTC in outcome prediction of mNPC patients will be uncovered.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiologically confirmed nasopharyngeal non-keratinizing carcinoma (WHO II, III).
* NPC patients with distant metastasis including synchronous distant metastasis at diagnosis and metachronous distant metastasis after radical treatment.
* A Karnofsky performance status score more than 70.
* The participants provided written informed consent.

Exclusion Criteria:

* A history of previous or synchronous malignant tumors.
* Suffering from severe mental illness synchronously.
* Suffering from severe heart or lung diseases.
* Obvious abnormality in liver and renal function.
* Women in pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NPC patients with distant metastasis
Sampling Method: Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 3 years

SECONDARY OUTCOMES:
The proportion of positives that are correctly identified as such | 3 years
  number of true positives divided by (number of true positives plus number of false negatives)
The proportion of negatives that are correctly identified as such | 3 years
  number of true negatives divided by (number of true negatives plus number of false positives)
The proportions of positive results in statistics and diagnostic tests that are true positive results. | 3 years
  number of true positives divided by number of positive calls
The proportions of negative results in statistics and diagnostic tests that are true negative results. | 3 years
  number of true negatives divided by number of negative calls

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Principal Investigator — Sun Yat-sen University

REFERENCES:
- [Result] Smerage JB, Barlow WE, Hortobagyi GN, Winer EP, Leyland-Jones B, Srkalovic G, Tejwani S, Schott AF, O'Rourke MA, Lew DL, Doyle GV, Gralow JR, Livingston RB, Hayes DF. Circulating tumor cells and response to chemotherapy in metastatic breast cancer: SWOG S0500. J Clin Oncol. 2014 Nov 1;32(31):3483-9. doi: 10.1200/JCO.2014.56.2561. Epub 2014 Jun 2. PMID 24888818
- [Result] Zhang Z, Shiratsuchi H, Lin J, Chen G, Reddy RM, Azizi E, Fouladdel S, Chang AC, Lin L, Jiang H, Waghray M, Luker G, Simeone DM, Wicha MS, Beer DG, Ramnath N, Nagrath S. Expansion of CTCs from early stage lung cancer patients using a microfluidic co-culture model. Oncotarget. 2014 Dec 15;5(23):12383-97. doi: 10.18632/oncotarget.2592. PMID 25474037
- [Result] Cristofanilli M, Hayes DF, Budd GT, Ellis MJ, Stopeck A, Reuben JM, Doyle GV, Matera J, Allard WJ, Miller MC, Fritsche HA, Hortobagyi GN, Terstappen LW. Circulating tumor cells: a novel prognostic factor for newly diagnosed metastatic breast cancer. J Clin Oncol. 2005 Mar 1;23(7):1420-30. doi: 10.1200/JCO.2005.08.140. PMID 15735118